CLINICAL TRIAL: NCT04813835
Title: Cognitive, Sleep, Neurophysiological Markers Among Suicidal Depressed Patients
Brief Title: Cognition, Sleep, Neurophysiology of Suicidal Depressed Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, waleed ashraf hamdy ahmed, Principal Investigator, Assiut University
Other Study IDs: cognition Suicidal Depression
Record Dates: First submitted 2021-02-26; First posted 2021-03-24 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Suicidal Depression
Keywords: cognition; sleep; neurophysiology; suicidal depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- suicidal depressed patients: psychiatric history suicidal scale mental state examination screening for sleep disturbance electroencephalography
- depressed patients: psychiatric history suicidal scale mental state examination screening for sleep disturbance electroencephalography
- control: psychiatric history suicidal scale mental state examination screening for sleep disturbance electroencephalography

SUMMARY:
evaluation whether suicidal major depressive disorder patients show a specific pattern of cognitive, sleep and neurophysiologic impairment as compared to non- suicidal major depressive disorder patient, and studying the correlation between the cognitive impairment, the sleep disturbance and the neurophysiologic impairment and suicidal behaviour Studying the cognitive profile in suicidal patient including studying, Comprehension, Attention, language production, reasoning, problem solving and decision making

DETAILED DESCRIPTION:
Suicide defined as when a person killing himself directly or indirectly act, with knowing that will produce this result carried out by the victim himself .Suicide is 14th leading cause of death worldwide, responsible for 1.5% of all mortality .suicide is the cause of death most directly affected by psychological factors. There is other stressors such as financial troubles, poverty, unemployment, homelessness and war may cause suicide. About (15-40%) of people leave a suicide note. Genetics appear to account for between 38% and 55% of suicidal behaviors . Suicide rates differ significantly between countries and over time. Percentage of death in 2013 in Africa was 1% Canada 11.1% china 12.7% India 23.2% and united states 14%. suicide is ranked as 10th leading cause of death in the united states. In china suicide is 5th leading cause of death.

Of all the psychiatric disorders. major depressive disorder in associated with the highest life time risk of suicide attempt and completion. Indeed. the life time risk of completing suicide in patient with (MDD) range from (35- 40 %, )in the world. Also in patient of mood disorder (MD) range about (8-15 %) of patient attempt suicide In an suicide attempt must be understand how and why some people's thought process lead them to decide to end their lives, there is several different cognitive impairment factors that seem to increase the risk of suicidal behavior such as cognitive rigidity, thought suppression. Agitation. Future thinking and goal adjustment .

Finding from studies in which behavioral test of cognitive rigidity are administrated to suicide attempter and clinical controls have support this notion.

studies illustrate the importance of control the sleep disorders as there is relationship between sleep disorders and suicidal behavior and subsequent suicidal thoughts and either self-harm behaviors or suicide attempt after controlling depressive symptoms Some studies have shown neurophysiologic aspects of suicidal behavior. An attempt has been made to reveal a correlation of results obtained in calculating the entropy and information Saturation of EEG with signs of dysontogenesis in patients with depression with- or without suicidal signs

ELIGIBILITY:
Inclusion Criteria:I) patients

a. Inclusion criteria:

1. Suicidal attempters, suicidal ideators, non-suicidal depressed were all diagnosed with major depression, or Bipolar disorder (BD) (depressive phase) by statistical manual of mental disorders. Patients meeting DSM-5 criteria. (APA-2013)
2. all participant provided written informed consent
3. age group above 18 years old II) control a. Inclusion criteria:

1. Match with the subjects in age group "above 18 years old" 2.no history of suicide attempt or ideation 3. no history of psychiatric disorder

Exclusion Criteria:

1. other psychiatric disorders
2. electroconvulsive therapy in the Previous six months
3. Neurologic disorders including stroke, epilepsy, brain injury and sensory disorders that precluded participating in cognitive assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: study population are grouped to 3 groups
  1. suicidal depressed patient
  2. depressed patients
  3. control or normal people
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Cognition among Suicidal Depressed patients | one day
  1. to determine the cognitive impairment among depressed suicidal patient compared to not depressed persons and to depressed non suicidal patients by 1-Mini-mental state examination: It as a basic tool used to assess the cognitive function; it includes tests of orientation, attention, memory, language and visual-spatial skills
  2. Montreal cognitive assessment scale:
  The test is a one-page 30-point test administered in approximately 10 minutes. Each participant had the test individually. it was used to assess several domains of cognition such as the short term memory recall task (5 points) involves two learning trials of five nouns and delayed recall after approximately 5minutes
sleep among Suicidal Depressed patients | 10 minutes
  Epworth sleepiness scale:
  The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness that is measured by use of a very short questionnaire. This can be helpful in screening of sleep disorders.
neurophysiological marker among Suicidal Depressed patients | 1 hour
  Standard Electroencephalogram "EEG":
  Conventional EEG will be done using the 8 channels Nihon Kohden machine '4217' employing scalp electrodes placed according to the international 10-20 system with bipolar and referential montages . for evaluation of power in alpha band

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F. Abd-ElAal, Professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] W. S. F. Pickering; Geoffrey Walford (2000). Durkheim's Suicide: a century of research and debate. Psychology Press. p. 25.
- [Background] Hassan, Wageeh .A.N., Noamany, M.M.(2020). . A clinical study of suicide in patients admitted in psychiatry unit in Assiut University. Middle East Current Psychiatry 27, 26